CLINICAL TRIAL: NCT03553329
Title: Study of the Variations of Albumin Level for Patients With Unresecable Stage IIIc or Stage IV Melanoma Treated by Anti BRAF and Anti MEK
Acronym: SVALMEL
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SVALMEL
Record Dates: First submitted 2018-04-03; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Unresecable Stage IIIc or IV Melanoma
MeSH Terms: interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dabrafenib — Monthly biological assessment which included: blood count, a blood electrolytes, an creatininemia, a dosage of urea, a dosage of transaminases, of gammaGT, of phosphatases alkaline, of LDH and of albumin.
  Other Names: trametinib

SUMMARY:
The therapeutic arsenal of metastatic melanoma has changed considerably over the past 10 years. The treatment of metastatic melanoma is now based on immunotherapy and targeted therapies, while the place of conventional chemotherapy becomes more restricted. Targeted therapies are indicated for BRAF mutated melanomas.

The mutation BRAF leads activation of MAP Kinases pathway and the proliferation of melanoma cell in the body . About 50% of metastatic melanoma is BRAF mutated. The most frequent mutation is the V600E. The targeted therapy by anti BRAF and anti MEK allows the double bloking of the MAP Kinases pathway. This treatment is more efficient than that of the anti BRAF alone. The association of anti BRAF and anti MEK have a global survival global rate of 41% at the 1 year, against 9% for the anti BRAF .

In 2014, a program of extended access to the association of anti BRAF and anti MEK (dabrafenib and trametinib) started in many french hospitals (Protocol Mekinist, Novartis laboratory). Patients who were included in this program and followed in Poitiers Hospital, had frequent abnormalities of albumin level without any sign of undernutrition.

Hypoabuminemia is a poor prognosis factor described in many cancers, including metastatic melanoma.

The only prognostic factor in metastatic melanoma is the rate of LDH . The level of albumin and its prognostic impact have not been studied for patients with a metastatic melanoma and treated by anti BRAF and anti MEK.

The objective of this studie was to analyze the variations of albumin level in patients with unresecable stage IIIc or stage IV melanoma treated in our Center by dabrafenib and trametinib

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans
* the patients with unresecable stage IIIc or IV melanoma with BRAF V600 E or K mutation,
* treated by dabrafenib and trametinib by the program of extended access (research protocol Mekinist)

Exclusion Criteria:

* Age < 18 ans
* patients who had less than 3 months of treatment,
* patients for which the albumin level could not be carried out before starting treatment, and after the first month

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable stage IIIc or stage IV melanoma, including the Mekinist research protocol
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Analyze the variations of albumin level in patients with unresecable stage IIIc or stage IV melanoma treated by dabrafenib and trametinib | 1 months
  Biological assessment
Analyze the variations of albumin level in patients with unresecable stage IIIc or stage IV melanoma treated by dabrafenib and trametinib | 3 months
  Biological assessment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU DE Poitiers, Poitiers, France